CLINICAL TRIAL: NCT02280148
Title: Accessing the Driving Skills After the Endoscopy of Intravenous Anesthesia by Driving Simulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhan yuanlin, Master of Beijing Friendship Hospital Gastroenterology, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BJFH-EC/2013-073
Record Dates: First submitted 2014-10-25; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Driving
Keywords: Propofol; gastroscopy and colonoscopy; driving simulator; driving ability; cognitive function; patients
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endoscopy of Intravenous Anesthesia (Experimental): 20-70 year-old volunteers who hold legitimate licenses were recruited to have gastroscopy or colonoscopy under intravenous anesthesia with propofol
  Interventions: Procedure: Endoscopy of Intravenous Anesthesia; Device: Driving Simulator; Drug: Propofol

INTERVENTIONS:
Procedure: Endoscopy of Intravenous Anesthesia — The dose of intravenous anesthesia drug and time was controlled by the anesthesiologist,endoscopists were responsible for gastroscopy or colonoscopy , nurses assisted endoscopists with biopsy.Each subject's initial dose of propofol were set at 2mg / kg, and were added properly by anesthesiologists additional according to the subjects' intraoperative sedation or surgical time.
Device: Driving Simulator
Drug: Propofol — 2mg / kg

SUMMARY:
The purpose of this study is to assess the driving and cognitive ability of gastrointestinal endoscopy patients at different time points after intravenous anesthesia (propofol for example), and to explore whether the driving and cognitive ability have a relationship with the blood concentration of propofol or not.

DETAILED DESCRIPTION:
20-70 year-old volunteers who hold legitimate licenses were recruited to have gastroscopy or colonoscopy under intravenous anesthesia with propofol, and before endoscopy using driving simulator and NCT to measure patients' driving ability and cognitive function as a baseline, in the same way, assessing patients' driving ability and cognitive function after 2h, 4h of the endoscopy , meantime collecting blood samples and separating blood plasma, using HPLC (High Performance Liquid Chromatography) to measure blood concentration of propofol.

ELIGIBILITY:
Inclusion Criteria:Outpatients who held a valid driver's license,were Aged 20 to 70 years old,had more than 2 years of driving experience, were with endoscopy or colonoscopy indications.

Exclusion Criteria:with gastroscopy or colonoscopy contraindications, long-term use of benzodiazepines or opioids,an American Society of Anesthesiologists physical status score (ASA) of Class IV or V,pregnant women,Emergency and hospitalized patients, allergy to narcotic drugs, with acute and chronic liver injury, have any clinical evidence of hepatic encephalopathy,severe based diseases and mental illness,serious adverse reactions such as dizziness, nausea, and vomiting in simulated driving.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
driving ability after of the endoscopy under Intravenous Anesthesia | within the first 4h after endoscopy
  before endoscopy using driving simulator to measure patients' driving ability as a baseline, in the same way, assessing patients' driving ability after 2h, 4h of the endoscopy.Driving simulation design scenes concluded low risk driving scene, medium risk driving scene and high risk driving scene.For low risk driving scene ,the observed indicators were average speed(m/s),average acceleration (m/s2), the average lane deviation (m), the maximum lane shift (m), the times of deviating from pathway .For medium risk driving scene ,the observed indicators were the minimum distance from overtaken vehicle, the times of overtaking intentions were observed in 80km/h and 40km/h speed limit.For high risk driving scene ,the observed indicators were maximum acceleration or deceleration, braking reaction time or accelerating reaction time.

SECONDARY OUTCOMES:
cognitive function after of the endoscopy under Intravenous Anesthesia | within the first 4h after endoscopy
  before endoscopy using NCT to measure patients'cognitive function as a baseline, in the same way, assessing patients'cognitive function after 2h, 4h of the endoscopy.common methods for assessing patients' cognitive function include MoCA Rating Scale (Montreal assessment)、MMSE (Mini-Mental State score), due to the poor reproducibility,neither of them were selected. NCT is usually used to diagnose and assess the progress of subclinical hepatic encephalopathy, this test is simple, reproducible, widely used to assess psychomotor functions recovery after anesthesia . NCT includes part A and B, in order to simplify ,only part A was used for the study.NCT-A requires participants line 1-25 numbers which were randomly distributed on paper in ascending order in time as short as possible, and their finish time will be recorded.

OTHER OUTCOMES:
measure blood concentration of propofol | within the first 4h after endoscopy
  collecting blood samples and separating blood plasma, using HPLC (High Performance Liquid Chromatography) to measure blood concentration of propofol after 2h,4h of endoscopy. Propofol blood concentration was measured by high performance liquid chromatography, which included high-performance liquid chromatography, C18 column, vortex mixer, high-speed centrifuges, reference reagents including propofol, thymol (internal standard) , methanol, acetonitrile, purified water, blank plasma. Measurement procedure can be summarized as the internal standard and plasma processing, the configuration of standard chromatographic conditions, HPLC analysis, the provision of the standard curve. The method detection limit was 0.5μg / ml, the scope of application of the linear concentration detection 0.5-4.0μg / ml. Determination of propofol blood concentration was done by researcher of Beijing Friendship Hospital drug testing experiment.

CONTACTS AND LOCATIONS:
Overall Officials: peng Li, doctor, Study Chair — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Riphaus A, Gstettenbauer T, Frenz MB, Wehrmann T. Quality of psychomotor recovery after propofol sedation for routine endoscopy: a randomized and controlled study. Endoscopy. 2006 Jul;38(7):677-83. doi: 10.1055/s-2006-925244. PMID 16810592
- [Derived] Hao XW, Zhan YL, Li P, Zhang ST, Yan XD, Li XM, Xiang W. Recovery of driving skills after endoscopy under propofol sedation: a prospective pilot study to assess the driving skills after endoscopic sedation using driving simulation. BMC Anesthesiol. 2023 Jun 24;23(1):223. doi: 10.1186/s12871-023-02122-z. PMID 37355565